CLINICAL TRIAL: NCT02418104
Title: A Randomized, Double-Blind, 2-Period Parallel-Arm Study to Assess the Immunogenicity of 2 Subcutaneous Doses of CHS-1701 (Coherus Pegfilgrastim) With 2 Subcutaneous Doses Neulasta® in Healthy Subjects
Brief Title: Assessing the Immunogenicity of 2 Subcutaneous Doses of CHS-1701 (Coherus Pegfilgrastim) With 2 Subcutaneous Doses Neulasta®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: CHS-1701-04
Record Dates: First submitted 2015-04-08; First posted 2015-04-16 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Immunity, Humoral
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHS-1701 (Experimental): CHS-1701 followed by CHS-1701
  Interventions: Drug: CHS-1701
- Neulasta (Active Comparator): Neulasta followed by Neulasta
  Interventions: Drug: Pegfilgrastim (Neulasta)

INTERVENTIONS:
Drug: CHS-1701
  Arms: CHS-1701
Drug: Pegfilgrastim (Neulasta)
  Other Names: Neulasta
  Arms: Neulasta

SUMMARY:
This is a randomized, double-blind, 2-period parallel study in healthy subjects to assess immunogenicity and safety of two sequential 6 mg subcutaneous (SC) injections of CHS-1701 compared with two sequential 6 mg SC injections of Neulasta®.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female of ages 18 to 50 inclusive
2. Body weight > 50 kg (110 lb.) and body mass index between 18 and 32 kg/m2 inclusive
3. Medically healthy with clinically insignificant findings based on medical history, 12-lead ECG, and physical examination
4. Negative urine pregnancy test in women of childbearing potential

Exclusion Criteria:

1. Previous exposure to pegfilgrastim or filgrastim, or known allergy to PEG (polyethylene glycol)
2. Chemistry and hematology values outside protocol specified range
3. Current or previous cancer, diabetes, or any clinically significant cardiovascular, metabolic, renal, hepatic, gastrointestinal, hematologic, respiratory, dermatological, neurological, psychiatric, or other disorder
4. History of chronic or acute respiratory illness within the past 4 weeks
5. Positive urine drug or alcohol screen or unwillingness to abstain from alcohol or recreational drugs for the duration of study participation
6. No prescription or nonprescription drugs during the study
7. Participation in an investigational clinical study within 30 days prior to screening
8. Known or suspected allergic reaction to latex

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 303 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To assess the immunogenicity of CHS-1701 compared to Neulasta | 84 days
  The primary objective of this study is to assess the immunogenicity of CHS-1701 compared to Neulasta based on the development of neutralizing antibodies (NAB) and the percent difference in ADA response

SECONDARY OUTCOMES:
Any potential impact of ADA or NAB on the pharmacokinetic (PK) profile of CHS-1701 using standard parameters (AUC, Cmax, ANCmax, or ANC (AUC0-t) | 84 days
Any potential impact of ADA or NAB on pharmacodynamic (PD) response as measured by absolute neutrophil count (ANC) | 84 days
Any potential impact of ADA or NAB on safety profile and tolerance of CHS-1701, as assessed by clinical adverse events (AEs), laboratory variables, vital signs, and local injection site reactions (ISRs) | 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Finck, MD, Study Director — Coherus Oncology, Inc.
Locations (4):
- United States (4):
  - Vince & Associates Clinical Research, Overland Park, Kansas
  - Medpace, Cincinnati, Ohio
  - ICON, San Antonio, Texas
  - Spaulding Clinical, West Bend, Wisconsin

REFERENCES:
- [Derived] Civoli F, Finck B, Tang H, Hodge J, O'Kelly H, Vexler V. Biosimilar Pegfilgrastim-cbqv Demonstrated Similar Immunogenicity to Pegfilgrastim in Healthy Subjects Across Three Randomized Clinical Studies. Adv Ther. 2022 Mar;39(3):1230-1246. doi: 10.1007/s12325-021-02024-x. Epub 2022 Jan 16. PMID 35034311